CLINICAL TRIAL: NCT06120543
Title: Correlation Between CYP1A2, ABCB1, CYP2C9 Gene Polymorphisms and Plasma Concentration of Agomelatine and Its Metabolites in Adult Patients With Depression
Brief Title: CYP1A2, ABCB1, CYP2C9 and Plasma Concentration of Agomelatine in Adult Patients With Depression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: wangqin01
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-08

CONDITIONS: Polymorphism, Genetic; Depression; CYP1A2 Polymorphism; CYP2C9 Polymorphism; Polymerase Chain Reaction; Plasma Concentration
Keywords: gene polymorphism; plasma concentration; agomelatine; adult depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 2ml of venous blood collected in ethylenediamine tetraacetic acid anticoagulant tubes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. The plasma concentrations of agomelatine and its two metabolites are simultaneously determined by High performance liquid chromatography-tandem mass spectrometry;
2. The gene polymorphisms of CYP1A2, ABCB1 and CYP2C9 are detected by fluorescence in situ hybridization or fluorescence polymerase chain reaction;
3. The correlation of CYP1A2, ABCB1, CYP2C9 gene polymorphisms with the blood concentration of agomelatine and its two metabolites is investigated by pharmacokinetic study;
4. According to the correlation between the above genotypes and blood drug concentration, a lean medication guidance scheme for agomelatine will be formed.

DETAILED DESCRIPTION:
1. research purpose and significance Through blood concentration monitoring, pharmacokinetics and gene detection technology, combined with clinical prospective research, the lean medication of agomelatine will be achieved. Objective to establish a method for analyzing the blood concentration of agomelatine and its two metabolites, which can be applied to routine detection in hospital. Objective to search for the genes related to the metabolism of agomelatine in vivo, and to detect the polymorphisms of related genes quickly and easily by fluorescence in situ hybridization or micro sequencing technology. Objective to explore the correlation between gene polymorphism and blood concentration of agomelatine and its two metabolites, and to make reasonable pharmaceutical recommendations for clinical lean drug use.
2. research content and design The plasma concentrations of agomelatine and its two metabolites are simultaneously detected by High performance liquid chromatography-tandem mass spectrometry; The gene polymorphisms of CYP1A2, ABCB1 and CYP2C9 are detected by fluorescence in situ hybridization or microsequencing; Objective to explore the correlation between CYP1A2, ABCB1, CYP2C9 gene polymorphisms and the blood concentration of agomelatine and its two metabolites by pharmacokinetic study.
3. research object

50 adult depression patients taking agomelatine

4 research steps

1. The plasma concentrations of agomelatine and its two metabolites are simultaneously detected by High performance liquid chromatography-tandem mass spectrometry;
2. The gene polymorphisms of CYP1A2, ABCB1 and CYP2C9 are detected by fluorescence in situ hybridization or fluorescence polymerase chain reaction;
3. The correlation of CYP1A2, ABCB1, CYP2C9 gene polymorphisms with the blood concentration of agomelatine and its two metabolites is investigated by pharmacokinetic study;
4. According to the correlation between the above genotypes and blood drug concentration, a lean medication guidance scheme for agomelatine will be formed.

5 evaluation index

1. The blood drug concentration monitoring method should have a certain degree of precision and accuracy, and meet the relevant requirements of the Chinese Pharmacopoeia; The gene detection method is required to be fast and simple, and the internal and external quality control should be carried out;
2. The medical record data should be collected completely, the privacy of patients should be respected, and the blood sample storage should meet the relevant conditions through the review of the hospital ethics committee;
3. The refined medication guidance scheme of agomelatine can be formed based on the data of therapeutic drug monitoring, gene detection and clinical research.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of depression; Sleep disorder.

Exclusion Criteria:

Mental disorder; Intelligence disorder; Dementia; Aphasia; Dysarthria; Consciousness disorder; Severe heart, kidney or liver dysfunction; Pregnant and lactating women; Malignant tumor.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult depression patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of Agomelatine | 3 hours after the patients take agomelatine
  Plasma concentration of Agomelatine
CYP1A2, ABCB1, and CYP2C9 genotypes | 3 hours after the patients take agomelatine
  CYP1A2, ABCB1, and CYP2C9 gene polymorphism
Plasma concentration of Agomelatine metabolites | 3 hours after the patients take agomelatine
  Plasma concentration of Agomelatine metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Qin Wang, Study Director — Affiliated Hospital of Nantong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maddukuri RK, Hema C, Sri Tejaswi K, Venkata Mounika M, Vegesana BP. Antidepressant efficacy of Agomelatine: Meta-analysis of placebo controlled and active comparator studies. Asian J Psychiatr. 2021 Nov;65:102866. doi: 10.1016/j.ajp.2021.102866. Epub 2021 Sep 20. PMID 34592623
- [Background] Arango C, Buitelaar JK, Fegert JM, Olivier V, Penelaud PF, Marx U, Chimits D, Falissard B; study investigators. Safety and efficacy of agomelatine in children and adolescents with major depressive disorder receiving psychosocial counselling: a double-blind, randomised, controlled, phase 3 trial in nine countries. Lancet Psychiatry. 2022 Feb;9(2):113-124. doi: 10.1016/S2215-0366(21)00390-4. Epub 2021 Dec 14. PMID 34919834
- [Background] Konstantakopoulos G, Dimitrakopoulos S, Michalopoulou PG. The preclinical discovery and development of agomelatine for the treatment of depression. Expert Opin Drug Discov. 2020 Oct;15(10):1121-1132. doi: 10.1080/17460441.2020.1781087. Epub 2020 Jun 22. PMID 32568567
- [Background] San L, Arranz B. Agomelatine: a novel mechanism of antidepressant action involving the melatonergic and the serotonergic system. Eur Psychiatry. 2008 Sep;23(6):396-402. doi: 10.1016/j.eurpsy.2008.04.002. Epub 2008 Jun 25. PMID 18583104
- [Result] Saiz-Rodriguez M, Ochoa D, Belmonte C, Roman M, Vieira de Lara D, Zubiaur P, Koller D, Mejia G, Abad-Santos F. Polymorphisms in CYP1A2, CYP2C9 and ABCB1 affect agomelatine pharmacokinetics. J Psychopharmacol. 2019 Apr;33(4):522-531. doi: 10.1177/0269881119827959. Epub 2019 Feb 21. PMID 30789308
- [Result] Guardiola-Lemaitre B, De Bodinat C, Delagrange P, Millan MJ, Munoz C, Mocaer E. Agomelatine: mechanism of action and pharmacological profile in relation to antidepressant properties. Br J Pharmacol. 2014 Aug;171(15):3604-19. doi: 10.1111/bph.12720. PMID 24724693
- [Result] Li M, Tang F, Xie F, Lv Y, Yu P, Liu Z, Cheng Z. Development and validation a LC-MS/MS method for the simultaneous determination of agomelatine and its metabolites, 7-desmethyl-agomelatine and 3-hydroxy-agomelatine in human plasma: Application to a bioequivalence study. J Chromatogr B Analyt Technol Biomed Life Sci. 2015 Oct 15;1003:60-6. doi: 10.1016/j.jchromb.2015.09.018. Epub 2015 Sep 18. PMID 26409931
- [Result] Xie F, Vermeulen A, Colin P, Cheng Z. A semiphysiological population pharmacokinetic model of agomelatine and its metabolites in Chinese healthy volunteers. Br J Clin Pharmacol. 2019 May;85(5):1003-1014. doi: 10.1111/bcp.13902. Epub 2019 Mar 21. PMID 30761579
- [Result] El-Deen AK, Magdy G, Shimizu K. A reverse micelle-mediated dispersive liquid-liquid microextraction coupled to high-performance liquid chromatography for the simultaneous determination of agomelatine and venlafaxine in pharmaceuticals and human plasma. J Chromatogr A. 2023 Nov 8;1710:464441. doi: 10.1016/j.chroma.2023.464441. Epub 2023 Oct 10. PMID 37832460
- [Result] Zhang H, Pu C, Wang Q, Tan X, Gou J, He H, Zhang Y, Yin T, Wang Y, Tang X. Physicochemical Characterization and Pharmacokinetics of Agomelatine-Loaded PLGA Microspheres for Intramuscular Injection. Pharm Res. 2018 Nov 8;36(1):9. doi: 10.1007/s11095-018-2538-7. PMID 30411255